CLINICAL TRIAL: NCT02541292
Title: Muscle Inflammation and Fat Infiltration in Patients Affected by FSHD
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Rigshospitalet, Denmark (Other)
Responsible Party: Principal Investigator, Julia Dahlqvist, MD, MD, Rigshospitalet, Denmark
Other Study IDs: H-15009760
Record Dates: First submitted 2015-09-02; First posted 2015-09-04 (Estimated); Last update posted 2018-09-04 (Actual); Status verified 2018-08

CONDITIONS: Facioscapulohumeral Muscular Dystrophy 1a
MeSH Terms: conditions — Facioscapulohumeral muscular dystrophy 1a

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Patient group: Patients over 18 years old with confirmed FSHD (facioscapulohumeral muscular dystrophy).
  Interventions: Other: No intervention, observational

INTERVENTIONS:
Other: No intervention, observational

SUMMARY:
Facioscapulohumeral muscular dystrophy (FSHD) is the second most common muscular dystrophy with approximately 500 patients in Denmark. It is characterized by weakness and wasting of the facial muscles, the muscles in the shoulder region and of the legs.

The primary aim of this study is to investigate possible links and order between inflammation and fat infiltration in the muscles in patients with FSHD.

Approximately 15 patients with FSHD will be recruited for repeated MRI-scans during a year where the inflammation and fat infiltration in the muscles can be quantified.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed FSHD

Exclusion Criteria:

* All contraindications for undergoing an MRI scan

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Persons in Denmark diagnosed with FSHD is invited to the study.
Sampling Method: Non-Probability Sample
Enrollment: 10 (Actual)
Dates: Start 2016-02; Primary Completion 2018-11 (Estimated); Study Completion 2018-11 (Estimated)

PRIMARY OUTCOMES:
Muscle inflammation | One MRI scan per subject (exam lasts approximately 60 min.)
  MRI (t2 mapping) will be used to quantify the inflammation in skeletal muscle.
Muscle fat fraction | One MRI scan per subject (exam lasts approximately 60 min.)
  The Dixon MRI will be used to quantify the fat fraction in skeletal muscle.

SECONDARY OUTCOMES:
Muscle strength | One muscle strength test per subject (exam lasts approximately 60 min.)
  Isokinetic muscle dynamometry will be used to measure muscle strength.

CONTACTS AND LOCATIONS:
Locations (1):
- Copenhagen Neuromuscular Center, Copenhagen, Denmark